CLINICAL TRIAL: NCT00735241
Title: Pilot Study of FOLFOX6 Plus Sir-Spheres® Microspheres (Chemo-radiotherapy) in Combination With Bevacizumab (Avastin) as a First Line Treatment in Patients With Nonresectable Liver Metastases From Primary Colorectal Carcinoma
Brief Title: FOLFOX6 Plus Sir-Spheres Microspheres Plus Avastin in Patients With Nonresectable Liver Metastases From Colorectal Carcinoma
Acronym: FAST
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Withdrawn by the study sponsor.
Sponsor: Sirtex Medical (Industry)
Responsible Party: David Cade, MD, Medical Director, Sirtex Technology Pty Ltd
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STX0207
Record Dates: First submitted 2008-08-13; First posted 2008-08-14 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Carcinoma; Liver Metastases
Keywords: colon cancer; colorectal cancer; liver metastases; SIR-Spheres Microspheres; yttrium-90; FOLFOX; Bevacizumab; chemo-radiation
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SIR-Spheres microspheres — SIR-Spheres yttrium-90 microspheres
Drug: FOLFOX6 cycles 1-3 — Oxaliplatin 60 mg/m2, IV infusion, q 2 weeks Leucovorin 200 mg/m2, IV infusion, q 2 weeks 5-Fluorouracil 400 mg/m2, IV bolus, q 2 weeks 5-Fluorouracil 2.4 g/m2, IV infusion, q 2 weeks
  Other Names: Eloxatin; Folinic acid; 5-FU
Drug: FOLFOX6 cycles 4 onwards — Oxaliplatin 85 mg/m2 given, IV infusion, q 2 weeks Leucovorin 200 mg/m2 given, IV infusion, q 2 weeks 5-Fluorouracil 400 mg/m2, IV bolus, q 2 weeks 5-Fluorouracil 2.4 g/m2, IV infusion, q 2 weeks
  Other Names: Eloxatin; Folinic acid; 5-FU
Drug: Bevacizumab cycles 3 onwards — Bevacizumab 10 mg/m2, IV infusion, q 2 weeks commencing with the third cycle of chemotherapy
  Other Names: Avastin

SUMMARY:
This pilot study will evaluate the safety and effectiveness of chemo-radiotherapy comprising a regimen of FOLFOX6 chemotherapy plus SIR-Spheres yttrium-90 microspheres (chemo-radiotherapy, also known as "chemo-SIRT"), in combination with the biologic therapy Bevacizumab (Avastin), for the first-line treatment of patients with liver metastases from colorectal carcinoma in whom surgical resection is not feasible.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum.
* Unequivocal and measurable CT evidence of liver metastases which are not treatable by surgical resection or local ablation with curative intent.
* ECOG performance status 0 - 1.
* Adequate hematological, renal and hepatic function.

Exclusion Criteria:

* Evidence of ascites, cirrhosis, portal hypertension, main portal vein tumor involvement or thrombosis as determined by clinical or radiologic assessment.
* Any extra-hepatic metastases other than metastases in the lungs and/or bones and/or abdominal or hilar lymph nodes. Central nervous system (CNS) metastases are not allowed.
* Previous radiotherapy delivered to the upper abdomen.
* Peripheral neuropathy > grade 1 (NCI-CTCv3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity and safety | from study entry until 28 days after last cycle of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Carter, MD, Principal Investigator — Rocky Mountain Cancer Center; Charlie Nutting, DO, Principal Investigator — Skye Ridge Medical Center
Locations (3):
- United States (3):
  - William Beaumont Hospital, Royal Oak, Michigan
  - Carolinas Medical Center, Charlotte, North Carolina
  - Sacred Heart Medical Center, Spokane, Washington